CLINICAL TRIAL: NCT04781621
Title: Foundational Ingredients of Robotic Gait Training for People with Spinal Cord Injury During Inpatient Therapy
Acronym: FIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chad Swank, Principal Investigator, Baylor Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSWRI IRB 020-483
Record Dates: First submitted 2021-02-03; First posted 2021-03-04 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-09

CONDITIONS: Spinal Cord Injuries
Keywords: Gait Training; Exoskeleton; Physical Therapy; Physical Rehabilitation and Medicine; Inpatient Rehabilitation; Robotic Gait Training; Randomized Control Trial
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Braces

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial. Patients are randomized into one of two groups: robotic exoskeleton gait training and usual care gait training.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Robotic Gait Training (Experimental): Patients in the Robotic Gait Training (RGT) group will receive 90 minutes per week of RGT once patients are deemed clinically appropriate as defined by being able to tolerate standing for 15 minutes without orthostatic intolerance. The duration of treatment will span the patient's length of stay in inpatient rehabilitation. The Ekso Bionics Ekso GT™ robotic exoskeleton will be used for RGT.
  Interventions: Device: Robotic Gait Training
- Usual Care Gait Training (Active Comparator): Usual Care (UC) gait training including body weight-supported treadmill training (BWSTT) and conventional overground walking.
  Interventions: Other: Usual Care Gait Training

INTERVENTIONS:
Device: Robotic Gait Training — Participants will wear an exoskeleton suit and receive robotic gait training with a physical therapist for 90 minutes each week. Robot gait training will include standing and walking activities while wearing the The Ekso Bionics Ekso GT™ robotic exoskeleton. Participants will be asked to complete questionnaires about walking and function. They will also be asked to wear a watch measuring their heart rate monitor.
  Other Names: EksoGT™ robotic exoskeleton
  Arms: Robotic Gait Training
Other: Usual Care Gait Training — Participants receive usual care gait training with a physical therapist for 90 minutes each week. Usual care gait training includes standard gait training involving standing and walking activities such as conventional overground walking, body weight-supported treadmill training (BWSTT), overground body weight-supported overground system, and various assistive devices (e.g., BWSTT, overground with braces, walker, etc.). Participants will be asked to complete questionnaires about walking and function. They will also be asked to wear a watch measuring their heart rate monitor and number of steps.
  Other Names: Standard of Care Gait Training; body-weight support treadmill training (BWSTT); Overground gait training with braces,
  Arms: Usual Care Gait Training

SUMMARY:
The FIRST project compares the dose of robotic gait training (RGT) with usual care gait training for patients with spinal cord injury (SCI) undergoing rehabilitation at Baylor Scott & White Institute for Rehabilitation (BSWIR).

DETAILED DESCRIPTION:
Spinal cord injury (SCI) due to trauma is estimated to affect 288,000 - 500,000 Americans, with about 17,700 new cases annually. Recovery of walking is a primary rehabilitation goal for patients and encouraged by therapists due to its relationship to quality of life, impact on health, psychological profile, and social participation after SCI. Recent technological advances with exoskeleton devices specifically for gait training may yield better walking recovery outcomes compared with usual care intervention approaches, such as body-weight support treadmill training (BWSTT) and overground gait training with braces, yet limited evidence exists for those with SCI.

Aim 1: Use a Community-Based Participatory Research approach to develop an robotic gait training (RGT) program that meets the unique needs of people after incomplete SCI during inpatient rehabilitation. This will be achieved by establishing and engaging an Advisory Board of key stakeholders to review evidence-based literature, advise the research team on the unique aspects and goals of inpatient rehabilitation for people with SCI, review the RGT, and make recommendations for amendments to the RGT program based on our interim and final outcomes of the study over the funding period.

Aim 2: Prospectively examine the efficacy of RGT compared to usual care gait training during inpatient rehabilitation in people with incomplete SCI.

Aim 3: Compare the intensity of RGT and usual care gait training during inpatient rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* 16 - 85 Years of Age
* All types of incomplete Spinal Cord Injury (SCI) (traumatic and non-traumatic)
* Acute/Subacute phase of recovery
* Medically stable as deemed by physician
* Undergoing medical care and inpatient rehabilitation at BSW
* Both genders and all races and ethnicities
* Meet the Ekso robotic exoskeleton frame limitations
* Continence of or a program for bladder and bowel management

Exclusion Criteria

* Moderate to Severe Traumatic Brain Injury (TBI)
* Degenerative diagnoses
* Wound located in proximity to the exoskeleton frame
* Severe osteoporosis/-penia as shown with dual energy x-ray absorptiometry (DXA)
* Pre-morbid developmental disability, significant psychological diagnosis, or other cognitive impairment

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Walking Index for Spinal Cord Injury - II (WISCI-II) | Within one week before discharge
  WISCI-II defines the physical limitation for gait secondary to impairment at the person level and indicates the ability of a person to walk after SCI. WISC-II rank orders the ability a person to walk on a scale of 0-20 with 0 representing no ability to stand or participate in assisted walking and 20 representing an ability to walk 10 meters with no devices, no braces, and no physical assistance.

SECONDARY OUTCOMES:
Gait speed via 10-Meter Walk Test (10MWT) | Within one week of admission before start of treatment; Within one week before discharge
  The 10MWT assesses gait speed (m/s) over a short duration.
Spinal Cord Independence Measure (SCIM) | Within one week of admission before start of treatment; Within one week before discharge
  The SCIM assesses self-care management, respiration and sphincter management, and functional mobility after a SCI. SCIM is composed of 19 items with total SCIM scores ranging from 0 (required assistance) to 100 (independence).
Numerical Pain Rating Scale (NPRS) | Within one week of admission before start of treatment; Within one week before discharge
  Pain is a significant problem in many individuals with SCI. A 0-10 Point Numerical Pain Rating Scale (NRS) is recommended as the outcome measure for pain intensity after SCI during acute and subacute phases. Pain severity can be categorized into 3 distinct groups as relates to pain interference: 1-3 (mild), 4-7 (moderate), 8-10 (severe).
Fatigue Severity Scale (FSS) | Within one week of admission before start of treatment; Within one week before discharge
  The Fatigue Severity Scale (FSS) is used to measure fatigue in neurologic disorders and measures the effects of fatigue on function. It is measure on the following scale:
  1. - Strongly Disagree
  2. - Disagree
  3. - Slightly Disagree
  4. - Neutral
  5. - Slightly Agree
  6. - Agree
  7. - Strongly Agree
Penn Spasm Frequency Scale (PSFS) | Within one week of admission before start of treatment; Within one week before discharge
  The PSFS is a self-report measure to assess a patient's perception of spasticity frequency and severity following a SCI. With excellent internal consistency (ICC = 0.90), the current version was modified from the original to include both frequency and severity.
Patient Health Questionnaire - 9 (PHQ-9) | Within one week of admission before start of treatment; Within one week before discharge
  The PHQ-9 is a self-report measure to assess the presence and intensity of depressive symptoms. For SCI, the PHQ-9 demonstrates excellent internal consistency (Chronbach's alpha = 0.87) and construct validity (r = 0.78).
General Anxiety Disorder (GAD-7) | Within one week of admission before start of treatment; Within one week before discharge
  The GAD-7 is a self-report measure to assess the presence of anxiety. Each items is scored on the following scale:
  0 - not at all
  1. - several days
  2. - more than half the days
  3. - nearly daily Total scores are calculated by adding all the score and provides a possible score cutoffs for 5 (mild anxiety), 10 (moderate anxiety) and 15 (severe anxiety).
International Spinal Cord Injury Quality of Life Basic Data Set | Within one week of admission before start of treatment; Within one week before discharge
  The International Spinal Cord Injury Quality of Life Basic Data Set is a three-item quality of life questionnaire suitable for SCI populations containing items assessing general life satisfaction, satisfaction with physical health, and satisfaction with psychological health. Items are answered on a 10-point likert scale that ranges from 0 (completely dissatisfied) to 10 (very satisfied).
Heart Rate (HR) | Immediately following every treatment until discharge, an average of 28 days
  Polar heart rate monitor (Polar® Unite) will provide data on the day, duration, and intensity (average and maximum) of gait training sessions for both RGT and UC. Participants will be provided a Polar heart rate monitor to wear during each gait training session for the entire length of the study, and gait training session data will be collected weekly. These monitors record beat to beat heart rates and store up to 16 sessions of heart rate data. Each week study staff will upload participants' heart rate data using Polar's FlowLink technology via the Polarpersonaltrainer.com website.
Ratings of Perceived Exertion (RPE) | Immediately following every treatment session until discharge, an average of 28 days
  The Borg RPE is a 15-point scale with verbal descriptors to standardize perceived exertion across tasks and individuals. Participants will be asked to provide a self-reported intensity level on the Borg Rating of Perceived Exertion Scale during RGT and UC gait training sessions. A self-report of 12 to 14 on the RPE indicates moderate intensity. The Borg RPE scale has been shown to be a valid measure of exercise intensity with weighted mean validity coefficient of 0.62 for HR.
Number of Steps | Immediately following every treatment session until discharge, an average of 28 days
  The Ekso device records several data points for each session including number of steps, "Up" time (the amount of time spent standing in the device), "Walk" time (the amount of time spent walking in the device), and device assistance scores. While all of these data values will be recorded to describe each RGT session and tracked to monitor progression of the RGT intervention, the number of steps per session will be utilized as an indicator of RGT session intensity.42,91 We will consult our Consumer Advocates for recommendations on incorporating device scores such as "Up" time and "Walk" time as additional measures of intensity.
  Number of steps for the UC group will be collected via pedometer during each gait training session. The number of steps captured on the device will be recorded on the case report form after each gait training session. The watch will be reset before each use.
Patient Perceptual Survey | Within one week before discharge
  This survey contains six open-ended questions assessing participant perception and satisfaction with treatment as well as asking participants to describe observable changes in functional activities.

CONTACTS AND LOCATIONS:
Overall Officials: Chad D Swank, PhD, Principal Investigator — Baylor Research Institute
Locations (1):
- Baylor Scott & White Institute for Rehabilitation, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swank C, Holden A, McDonald L, Driver S, Callender L, Bennett M, Sikka S. Foundational ingredients of robotic gait training for people with incomplete spinal cord injury during inpatient rehabilitation (FIRST): A randomized controlled trial protocol. PLoS One. 2022 May 10;17(5):e0267013. doi: 10.1371/journal.pone.0267013. eCollection 2022. PMID 35536844